CLINICAL TRIAL: NCT00442195
Title: Procurement and Analysis of Blood, Bone Marrow, and Buccal Mucosa Samples From Healthy Volunteers to Support Clinical and Translational Research Projects in the NHLBI
Brief Title: Collection and Analysis of Blood, Bone Marrow, and Buccal Mucosa Samples From Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070113; 07-H-0113
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12-04

CONDITIONS: Healthy Volunteers
Keywords: Tissue Procurement; Sample Collection; Biologic Samples; Laboratory Research Specimens; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy Volunteers

SUMMARY:
The Hematology Branch of the National Heart, Lung, and Blood Institute is doing a variety of laboratory research experiments that require blood and tissue samples from healthy volunteers. This protocol provides a mechanism for collecting these tissue samples. Research includes studies of normal and abnormal formation of blood cells, viral blood diseases, the role of the immune system in marrow failure and genetic risk factors for aplastic anemia.

Healthy normal volunteers 8 years of age and older may be eligible for this study. Samples are collected as follows:

* Blood samples: Participants 8 years of age and older donate up to 4 tablespoons of blood, which is obtained from a needle placed in an arm vein.
* Participants 8 years of age and older donate a buccal mucosa sample (cells from the inside of the cheek). The inside of the cheek is scraped gently with a nylon brush.
* Participants 18 years of age and older donate a bone marrow sample. The bone marrow is obtained from the hip bone. The skin over the area is wiped clean with alcohol and iodine, and then a local anesthetic is injected under the skin and also into the bone. When the area is numb, a bone marrow aspiration needle is introduced through the bone surface into the marrow. The marrow cells are collected using a syringe connected to the needle.

DETAILED DESCRIPTION:
The purpose of this protocol is to collect and analyze blood (ages 8 and older), bone marrow (ages 18 and older), skin tissue samples (ages 18 and older), and/or buccal mucosa samples (ages 8 and older) from healthy volunteers. Samples will be used for clinical and translational research in the NHLBI and are indispensable for many of our research projects, including studies of normal and abnormal hematopoiesis, the viral etiology of blood diseases, the role of the immune system in marrow failure and genetic risk factors for aplastic anemia. This protocol provides a mechanism for collection, tracking, storing, dispensing, analyzing and disposing of these laboratory research samples.

ELIGIBILITY:
* INCLUSION CRITERIA:

Self-declared healthy volunteer (for blood and buccal mucosa sample donors).

Be healthy, as determined by Principal Investigator or designee based on recent (<3 months) history, physical and laboratory results (for bone marrow and skin tissue sample donors).

<TAB><TAB><TAB><TAB><TAB>

Age 8 years and older (no upper limit) for blood and buccal mucosa sampling.

OR

Ages 18 years or older (no upper limit) for bone marrow or skin tissue sampling.

EXCLUSION CRITERIA:

Unable to comprehend the investigational nature of the protocol participation.

CBC determined outside expected normal ranges for the subject (bone marrow and skin tissue donors only).

Pregnancy

Age less than 18 years for skin tissue sampling, bone marrow aspirate and biopsy.

Off campus volunteers for skin tissue sampling bone marrow aspirate and biopsy.

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-03-03 (Actual)

PRIMARY OUTCOMES:
To obtain blood, bone marrow, and skin punch biopsy samples and/or buccal mucosa samples from subjects seeking to participate as healthy volunteers in NIH laboratory research studies. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Traba J, Kwarteng-Siaw M, Okoli TC, Li J, Huffstutler RD, Bray A, Waclawiw MA, Han K, Pelletier M, Sauve AA, Siegel RM, Sack MN. Fasting and refeeding differentially regulate NLRP3 inflammasome activation in human subjects. J Clin Invest. 2015 Nov 3;125(12):4592-600. doi: 10.1172/JCI83260. PMID 26529255
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2007-H-0113.html